CLINICAL TRIAL: NCT05279976
Title: The Effect of Visualized Education and Distraction in the Preoperative Process on Reducing the Anxiety of Children and Their Parents: a Randomized Controlled Study
Brief Title: Reducing the Anxiety of Children and Their Parents in the Preoperative Process
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Collaborators: Isparta University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Ayla Kaya, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AkdUniversity
Record Dates: First submitted 2022-02-23; First posted 2022-03-15 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Preoperative Care; Child; Parent; Anxiety
Keywords: Preoperative care; Child; Parents; Nursing; Randomized controlled trial
MeSH Terms: conditions — Anxiety Disorders | interventions — Osteogenesis, Distraction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Children receiving education-Intervention group 1 (35 children) (Experimental): Children in the intervention group 1 will be told by the researchers the operation preparation room and the pre-anesthesia process with a picture booklet. It will be ensured that the child and parent are together during the training. The booklet, which is printed separately for each child, will be given to the child and the parent after an average of 15-20 minutes of narration is completed. Simultaneous visual presentation will be made with the content of the picture booklet being explained to the child. While one of the researchers will explain the pre-operative process from the picture booklet, the other will explain the pre-operative preparation process simultaneously with the picture booklet by putting on the bonnet, mask and glove, and with the balloon inflated by the child. In this way, the pictures shown in the picture booklet will be matched with the real environment.
  Interventions: Other: Visualized Education
- Children who are distracted-Intervention group 2 (35 children) (Experimental): Children included in intervention group 2 will be given a kaleidoscope. Each child will be given a separate kaleidoscope. It will be ensured that the child is with the parent while the child is looking at the kaleidoscope for an average of 15-20 minutes. After the attempt is over, the kaleidoscope will be presented to the child.
  Usage of Kaleidoscope: It is a game tool that reproduces the outside image when viewed from inside the kaleidoscope. This image is obtained thanks to the glasses placed inside the kaleidoscope at different angles, and the images change as the kaleidoscope is rotated. Inside the kaleidoscope, there are mirrors or glasses placed with an inclination of 60 degrees. When viewed from one side of the kaleidoscope, images are often seen that are not the same.
  Interventions: Other: Distraction
- Control group of children (35 children) (No Intervention): After obtaining informed consent from the children and parents included in the control group after randomization, the pre-test (first measurement) will be applied. The final test (Second Measurement) will be applied immediately after the child wears the surgical gown.
- Parents of children receiving education-Intervention group 1 (35 parents) (Experimental): The parents of children included in intervention group 1 will also be in intervention group 1.It will be ensured that the child and parent are together during the training. The booklet, which is printed separately for each child, will be given to the child and the parent after an average of 15-20 minutes of narration is completed.
  Interventions: Other: Visualized Education
- Parents of distracted children-Intervention group 2 (35 parents) (Experimental): The parents of children included in intervention group 2 will also be in intervention group 2. Children included in intervention group 2 will be given a kaleidoscope. Each child will be given a separate kaleidoscope. It will be ensured that the child is with the parent while the child is looking at the kaleidoscope for an average of 15-20 minutes.
  Interventions: Other: Distraction
- Control group of parents (35 parents) (No Intervention): The parents of children included in control group will also be in control group.

INTERVENTIONS:
Other: Visualized Education — The child assigned to intervention group 1 will be told the operation preparation room and the pre-anesthesia process through the picture booklet prepared immediately after the pre-test (first measurement). Children included in this group will be provided to touch the bonnet, mask, gloves and self-inflated balloon (representing the ambu device), and the questions of the child and the parent will be answered.
  Arms: Children receiving education-Intervention group 1 (35 children); Parents of children receiving education-Intervention group 1 (35 parents)
Other: Distraction — Children included in intervention group 2 will be given a kaleidoscope. Each child will be given a separate kaleidoscope. It will be ensured that the child is with the parent while the child is looking at the kaleidoscope for an average of 15-20 minutes. After the attempt is over, the kaleidoscope will be presented to the child.
  Arms: Children who are distracted-Intervention group 2 (35 children); Parents of distracted children-Intervention group 2 (35 parents)

SUMMARY:
It is emphasized in the studies that the child and parent anxiety that occurs in pediatric surgery should be prevented or reduced. According to previous studies, one way to reduce child and parent anxiety in the preoperative process is to inform the child and family with preoperative family-centered activities. Teaching children anxiety coping skills with the involvement of their parents can reduce preoperative anxiety. This study was planned to evaluate the effect of visualized education and kaleidoscope distraction on children and parents' anxiety on the day of surgery in the preoperative period.

DETAILED DESCRIPTION:
Aim: This study was planned to evaluate the effect of visualized education and kaleidoscope distraction on children and parents' anxiety on the day of surgery in the preoperative period.

Method: This study was planned as a randomized controlled trial. The sample of the study will consist of 105 children aged 5-12, who will be operated on at Akdeniz University Hospital, and their parents. Randomization result; Education group=35, distraction group=35, and control group=35 children, a total of 105 children in 3 groups and their parents were planned to be included in the study. Child and parent information form will be used to collect data, Modified Yale Preoperative Anxiety Scale will be used to collect data in child sample, and Spielberger State Anxiety Scale will be used to collect data in parent sample.

Intervention and Data Collection: The study was planned to be implemented in the Akdeniz University Hospital Operating Room Patient Preparation Room, after the approval of the Akdeniz University Ethics Committee and the written permission of the Akdeniz University Hospital. It will be ensured that the child and parent are together during the initiatives. No intervention will be applied to the parents included in the sample of the study. After explaining the purpose of the study to the child and parent who agreed to participate in the study and obtaining consent, randomization will be performed. The child assigned to intervention group 1 will be told the operation preparation room and the pre-anesthesia process through the picture booklet prepared immediately after the pre-test (first measurement). Children included in this group will be provided to touch the bonnet, mask, gloves and self-inflated balloon (representing the ambu device), and the questions of the child and the parent will be answered. Children and parents included in this group will form intervention group 1 (35 children, 35 parents).

The child, who was assigned to intervention group 2 as a result of randomization, will be provided with the use of kaleidoscope, which is a distraction technique, immediately after the pre-test (first measurement). The second measurement will be made immediately after the child wears the surgical gown. Children and parents included in this group will form intervention group 2 (35 children, 35 parents).

Children randomized to the control group will not receive any intervention. A pre-test (first measurement) will be made for the child who is assigned to the control group as a result of randomization, and the second measurement will be made immediately after the child wears the surgical gown. Children and parents included in this group will form control group (35 children, 35 parents).

After all post-test (second measurement) applications are completed, the effectiveness of the interventions and their comparison with each other will be evaluated. After the post-test application of the research is completed, the data obtained will be analyzed using the Statistical Package of Social Science (SPSS) 23.0 software package program. The process of evaluating the data will be carried out with the support of a statistician.

ELIGIBILITY:
Inclusion Criteria:

* Being a child between the ages of 5-12 for which a surgical operation is planned
* Being the parent of a child between the ages of 5 and 12 whose surgical operation is planned
* Not having vision, hearing or speech problems
* Not have a mental or neurological disability
* Children and parents who can speak and understand Turkish will be included in the study.

Exclusion Criteria:

* Change in surgical operation date
* Using another distraction technique
* Children who do not arrive on the day of surgery will not be included in the study.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Children receiving education-Intervention group 1 | Anxiety levels of children during the preoperative period will be evaluated twice, in the operating room waiting room and immediately after the child wears the surgical gown. The second measure is the decrease in test scores, the outcome measure.
  The decrease in anxiety level of children in this group who received visualized education is a measure of outcome. This decrease will be measured by the "Modified Yale Preoperative Anxiety Scale". In the intervention group, the first (pre-test) measurement will be made in the operating room waiting room, and the second (post-test) measurement will be made with the same measuring instrument right after the surgical gown is put on. The scale consists of twenty-two items and five categories. Each category receives a score out of four. The higher the score on the scale, the greater the anxiety. In the post-test, it will be evaluated whether there is an decrease according to the pre-test score. If there is a decrease in the "posttest" scores compared to the "pretest" scores, it can be said that the visualized education has an positive effect on preoperative anxiety. Statistical significance will be set at p < 0.05.
Children who are distracted-Intervention group 2 | Anxiety levels of children during the preoperative period will be evaluated twice, in the operating room waiting room and immediately after the child wears the surgical gown. The second measure is the decrease in test scores, the outcome measure.
  The decrease in anxiety level of children in this group who are distracted by the keladoscope is a measure of outcome. This decrease will be measured by the "Modified Yale Preoperative Anxiety Scale". In the intervention group, the first (pre-test) measurement will be made in the operating room waiting room, and the second (post-test) measurement will be made with the same measuring instrument right after the surgical gown is put on. The scale consists of twenty-two items and five categories. Each category receives a score out of four. The higher the score on the scale, the greater the anxiety. In the post-test, it will be evaluated whether there is an decrease according to the pre-test score. If there is a decrease in the "posttest" scores compared to the "pretest" scores, it can be said that the distracted by the keladoscope has an positive effect on preoperative anxiety. Statistical significance will be set at p < 0.05.
Parents of children receiving education-Intervention group 1 | Anxiety levels of parents during the preoperative period will be evaluated twice, in the operating room waiting room and immediately after the child wears the surgical gown. The second measure is the decrease in test scores, the outcome measure.
  The decrease in anxiety level of parents in this group who parents of children receiving education is a measure of outcome. This decrease will be measured by the "Spielberger State Anxiety Scale". In the intervention group, the first (pre-test) measurement will be made in the operating room waiting room, and the second (post-test) measurement will be made with the same measuring instrument right after the child to be operated on is wearing a surgical gown. The 4-point Likert-type scale, consisting of 20 items in total, measures the anxiety of the person at a certain time. For scores above 42 points, it indicates a high level of anxiety. In the post-test, it will be evaluated whether there is an decrease according to the pre-test score. If there is a decrease in the "posttest" scores compared to the "pretest" scores, it can be said that the education has an positive effect on preoperative anxiety. Statistical significance will be set at p < 0.05.
Parents of distracted children-Intervention group 2 | Anxiety levels of parents during the preoperative period will be evaluated twice, in the operating room waiting room and immediately after the child wears the surgical gown. The second measure is the decrease in test scores, the outcome measure.
  The decrease in anxiety level of parents in this group who parents of distracted children is a measure of outcome. This decrease will be measured by the "Spielberger State Anxiety Scale". In the intervention group, the first (pre-test) measurement will be made in the operating room waiting room, and the second (post-test) measurement will be made with the same measuring instrument right after the child to be operated on is wearing a surgical gown. The 4-point Likert-type scale, consisting of 20 items in total, measures the anxiety of the person at a certain time. For scores above 42 points, it indicates a high level of anxiety. In the post-test, it will be evaluated whether there is an decrease according to the pre-test score. If there is a decrease in the "posttest" scores compared to the "pretest" scores, it can be said that distracted by the kaleidoscope has an positive effect on preoperative anxiety. Statistical significance will be set at p < 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Ayla Kaya, RN, PhD, Study Director — Akdeniz University Faculty of Nursing; Fahriye Pazarcıkcı, RN, PhD, Study Chair — Isparta University of Applied Sciences; Emine Efe, RN, PhD, Study Chair — Akdeniz University Faculty of Nursing
Locations (1):
- Akdeniz University, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aytekin A, Doru O, Kucukoglu S. The Effects of Distraction on Preoperative Anxiety Level in Children. J Perianesth Nurs. 2016 Feb;31(1):56-62. doi: 10.1016/j.jopan.2014.11.016. Epub 2015 Nov 11. PMID 26847781
- [Background] Baghele A, Dave N, Dias R, Shah H. Effect of preoperative education on anxiety in children undergoing day-care surgery. Indian J Anaesth. 2019 Jul;63(7):565-570. doi: 10.4103/ija.IJA_37_19. PMID 31391620
- [Background] Bulut M, Kucuk Alemdar D, Bulut A, Salci G. The Effect of Music Therapy, Hand Massage, and Kaleidoscope Usage on Postoperative Nausea and Vomiting, Pain, Fear, and Stress in Children: A Randomized Controlled Trial. J Perianesth Nurs. 2020 Dec;35(6):649-657. doi: 10.1016/j.jopan.2020.03.013. Epub 2020 Jul 20. PMID 32703758
- [Background] Dwairej DA, Obeidat HM, Aloweidi AS. Video game distraction and anesthesia mask practice reduces children's preoperative anxiety: A randomized clinical trial. J Spec Pediatr Nurs. 2020 Jan;25(1):e12272. doi: 10.1111/jspn.12272. Epub 2019 Oct 1. PMID 31576651
- [Background] Pazarcikci F, Efe E. Effect of care programme based on Comfort Theory on reducing parental anxiety in the paediatric day surgery: Randomised controlled trial. J Clin Nurs. 2022 Apr;31(7-8):922-934. doi: 10.1111/jocn.15945. Epub 2021 Jul 8. PMID 34240490 (Retraction: PMID 35429066 J Clin Nurs. 2022 Jun;31(11-12):1721)
- [Background] Stewart B, Cazzell MA, Pearcy T. Single-Blinded Randomized Controlled Study on Use of Interactive Distraction Versus Oral Midazolam to Reduce Pediatric Preoperative Anxiety, Emergence Delirium, and Postanesthesia Length of Stay. J Perianesth Nurs. 2019 Jun;34(3):567-575. doi: 10.1016/j.jopan.2018.08.004. Epub 2018 Nov 7. PMID 30413359